CLINICAL TRIAL: NCT06824831
Title: Analysis of the Effects Derived from the Use of Microporous Polysaccharide Hemospheres in Mastectomies with or Without Associated Lymphadenectomy
Brief Title: Use of Microporous Polysaccharide Hemispheres in Breast Cancer Patients Undergoing Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Marcos Adrianzén Vargas, Medical Doctor, Instituto de Investigacion Sanitaria INCLIVA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Arista_HCUV
Record Dates: First submitted 2025-01-25; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2022-06

CONDITIONS: Mastectomy; Lymphadenectomy; Breast Neoplasm Malignant Female; Breast Surgery; Seroma Following Procedure
Keywords: breast cancer; breast surgery; lymphadenectomy; seroma
MeSH Terms: conditions — Breast Neoplasms; Seroma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients receive microporous polysaccharide hemospheres (treatment arm) (Active Comparator)
  Interventions: Drug: Patients receive microporous polysaccharide hemospheres.
- Patients NOT receive microporous polysaccharide hemospheres (control arm) (Other)
  Interventions: Drug: Patients DO NOT receive microporous polysaccharide hemospheres.

INTERVENTIONS:
Drug: Patients receive microporous polysaccharide hemospheres. — Patients were randomized to receive microporous polysaccharide hemospheres, after mastectomy was done.
  Arms: Patients receive microporous polysaccharide hemospheres (treatment arm)
Drug: Patients DO NOT receive microporous polysaccharide hemospheres. — Patients were randomized to NOT receive microporous polysaccharide hemispheres after mastectomy was done.
  Arms: Patients NOT receive microporous polysaccharide hemospheres (control arm)

SUMMARY:
You should know that your participation in this study is voluntary and that you may decide NOT to participate. If you decide to participate, you may change your decision and withdraw your consent at any time, without altering your relationship with your physician or harming your health care.

The presence of seroma (accumulation of fluid in the surgical area) is a very common complication after mastectomy and axillary emptying, it can occur in up to 50% of cases. Its presence entails the need to wear a drain for days and causes numerous visits to the surgery office and/or emergency room for control of the drain itself or for puncture of the seroma that develops after removal of the drain.

The aim of the study is to assess whether the use of powdered hemostatics (microporous polysaccharide hemispheres whose commercial name is AristaTM) on the surgical bed reduces seroma formation after removal of the whole breast or all the fat in the axilla (mastectomy or axillary emptying). In the case of being able to demonstrate the benefits of its use, the discomfort of carrying an aspiration drain for a long time could be avoided, and the possibility of complications secondary to the use of the same could be reduced.

The main characteristics of the present study are:

* The total number of patients included in the study will be 120.
* The study will include all patients diagnosed with breast cancer in whom it is necessary to perform a mastectomy, whether or not associated with axillary emptying. If you are included in the study you may be included in one of the two groups (control group and study group). In the study group AristaTM will be used in the surgical bed after surgery, while in the control group AristaTM will not be used. In both groups, aspirative drains and chest bandage will be used after surgery.
* Assignment to one group or the other will take place at the time of surgery and will be randomized.
* The duration of the study will be until the total number of patients required is completed.
* The number of visits and controls will depend on the time it is necessary to carry the drainage or on the persistence of the seroma. It will not be different from the usual one in case you decide not to participate in the study.
* No additional tests or complementary explorations will be necessary for participating in the study. The only thing necessary will be the strict control of the daily debit accumulated in the drainage canister while you are carrying it, this control is also necessary and does not differ in case you decide not to participate in the study.

No additional risk is foreseen since no procedure outside the usual clinical practice is going to be performed.

You may not gain any health benefit from participating in this study, but you may help to learn about the usefulness of the AristaTM by avoiding the occurrence of seroma or the discomfort of wearing a drain for a long time in future patients requiring an intervention such as yours.

The data collected for the study will be identified by a code, so that it does not include information that can identify you, and only your study doctor/collaborators will be able to relate this data to you and your medical history. Therefore, your identity will not be disclosed to anyone except in the case of a medical emergency or legal requirement.

Access to your personally identifiable information will be restricted to the study physician/collaborators, competent authorities, the Research Ethics Committee and personnel authorized by the sponsor (study monitors, auditors), when required to verify the study data and procedures, but always maintaining the confidentiality of the same in accordance with current legislation.

If you decide to withdraw your consent to participate in this study, no new data will be added to the database, but the data already collected will be used.

In addition, you can limit the processing of data that are incorrect, request a copy or have the data you have provided for the study transferred to a third party (portability).

The encrypted data may be transmitted to third parties and other countries, but in no case will it contain information that can directly identify you, such as your first and last name, initials, address, social security number, etc. In the event that this transfer occurs, it will be for the same purposes of the study described or for use in scientific publications, but always maintaining the confidentiality of the same in accordance with current legislation.

Your participation in this study does NOT involve the collection and use of biological samples.

DETAILED DESCRIPTION:
INTRODUCTION Breast cancer is one of the most frequently diagnosed neoplasms worldwide. The global incidence of breast cancer has been increasing during the past decades. It was estimated to affect approximately 2.3 million women globally in 2020, causing about 685,000 deaths, and its incidence is likely to increase in the years to come.

Locoregional therapy includes surgery to remove the tumour, which remains one of the key interventions in the management of breast cancer. However, different postoperative complications can arise, especially when axillary surgery is concomitantly performed. Among these, seroma formation is one of the most common, with a described incidence of up to 90%, defined as an accumulation of serous fluid under the skin. Although seromas are not usually considered a serious complication, their appearance can result in wound infection and delayed wound healing and might delay adjuvant treatments.

Different strategies are currently available, such as wound drainage, external compression dressings, glues, and drugs, to reduce postoperative seroma formation. Several meta-analyses have evaluated the use of these techniques however, some of these studies have highlighted the lack of the overall quality of the reviewed data.

In this context, hemostatic agents have emerged as an alternative in surgical procedures. Among these, a powder composed of plant-based microporous polysaccharide hemospheres (MPH)11 has been approved as an adjunctive hemostatic device. MPH functions as a sieve absorbing fluid and concentrating clotting factors and is absorbed within 24 to 48 hours. Over a decade ago, MPH showed a significant reduction in seroma volume after mastectomy and axillary dissection in an animal model. In addition, these authors demonstrated a reduction in seroma's total protein, albumin and lactate dehydrogenase levels and white blood cell count in animals receiving MPH, suggesting a reduced seroma formation after MPH application. More recent studies conducted in patients undergoing different surgical interventions have evaluated the potential of MPH in postoperative seroma formation. However, data on MPH effectiveness in reducing seroma formation are heterogeneous.

Considering the above, the main goal of the study was to evaluate the use of MPH in reducing postoperative seroma formation in patients with breast cancer undergoing mastectomy with or without axillary lymphadenectomy.

In addition, we aimed to assess the emergence of immediate postoperative complications (first 72 hours) and the number of visits to the emergency department, to identify clinical factors associated with seroma formation, and to determine the relation between the amount of MPH and seroma formation, drain output, lymphadenectomy, and body mass index (BMI).

OBJECTIVE This study aimed to evaluate the effects of MPH in reducing postoperative seroma formation in patients undergoing mastectomy, with or without associated lymphadenectomy.

METHODS Study design and population This prospective, controlled study was conducted at the Hospital Clínico Universitario de Valencia between 2020 and 2022. All patients ≥18 years old diagnosed with breast cancer undergoing mastectomy with or without axillary lymphadenectomy were consecutively invited to participate in the study. No exclusion criteria were applied. Written informed consent was obtained before the inclusion. During the intraoperative period, patients were randomized 1:1 to receive microporous polysaccharide hemispheres (AristaTM AH; MPH treatment arm) or not (control arm). Management of postoperative complications in both groups followed routine clinical practice.

The study was approved by the Ethics Committee for Research of the Hospital Clínico Universitario de Valencia (code 2024/118) and developed following the ethical standards of the Helsinki Declaration of 1975.

Surgical procedure The surgical procedure followed the standard protocol for this type of intervention. In most cases, the Stewart incision was adapted according to the location of the tumour and/or the necessity for skin resection. The axillary approach, whether for the sentinel lymph node biopsy or in cases requiring an axillary dissection, was performed through the same incision used for the mastectomy. After the resection of the mammary gland and/or axillary node dissection, the area of the surgical site was measured. The area was calculated in all cases by measuring the length of the surgical site from medial to lateral and cranial to caudal, multiplying these dimensions to obtain the area in cm². Following the mastectomy and measurement of the surgical site, the patient was randomized. If assigned to the Arista group, the product was applied to cover the entire surface, and the amount used was recorded in grams. In all cases, suction drains were placed, and a compressive bandage was applied to all patients in both groups. They were discharged on the same day as the surgery and were followed up in outpatient clinics 24-48 hours post-operation. Each patient was provided with a sheet to record the daily drainage output. During follow-up visits, the drain was removed when the output was less than 30 ml over 24 hours, and patients were monitored until the complete resolution of the seroma. In cases where a seroma developed, drainage was performed via puncture and aspiration.

Study variables Sociodemographic (sex, age), clinical (weight, height, obesity, body mass index, diabetes, previous breast cancer and surgery, cardiopathy, hypertension, chronic obstructive pulmonary disease, smoking status, use of antiplatelet drugs and anticoagulants) and breast cancer-related (affected breast, inflammatory carcinoma, diagnostic, molecular determination, adjuvant treatment, sentinel node affectation) characteristics were collected before the procedure. Variables related to the surgical procedure (lymphadenectomy, mastectomy, surgical intervention time, surgical area, intraoperative complications, drainage, antibiotic prophylaxis, dressing, hemostasia, bleeding risk) and patient follow-up (surgical wound infection and dehiscence, seroma, time with drainage, volume of drain output, seroma punctures, postoperative complications, hematoma, follow-up time, outpatient visits, hospital length of stay, death) were also collected.

Sample size calculation The sample size was estimated based on data from a previous review in which the percentage of seromas in mastectomy after a drain insertion was 46.21%19.

To find as statistically significant a proportion difference of ≥25% between treatment and control arms (estimated at 0.2121 and 0.4621 for the MPH and control group, respectively) and accepting a confidence level of 5% (alpha risk) and a power of 80% (beta risk) in a two-tailed test, a total sample size of 116 patients (58 per treatment arm) was estimated. A drop-out rate of 5% was anticipated.

Statistical analysis Quantitative variables were presented as mean and standard deviation (SD). For qualitative variables, relative and absolute frequencies were calculated. The normality of data distribution was tested with the Shapiro-Wilk test.

The association between MPH and qualitative variables was assessed using the Chi-square or Fisher's exact test, while the association between MPH and quantitative variables was evaluated using Student's t-test or Mann-Whitney U test. A univariate logistic regression model was also used to quantify the association between seroma formation and the MPH treatment arm. Results were presented as Odds Ratio (OR) and 95% confidence interval (95% CI). To evaluate the association between the quantity (cm2/g) of MPH used during surgery and the drain output, Pearson's correlation coefficient or Spearman's non-parametric correlation coefficient were used.

All analyses were performed using the STATA v.14 software. A p-value < 0.05 was considered statistically significant for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) over 18 years of age.
* Patients diagnosed with breast cancer and scheduled for surgical treatment either simple mastectomy or mastectomy plus axillary mastectomy or mastectomy plus axillary emptying.
* Patients who sign the informed consent for mastectomy and/or mastectomy plus axillary emptying.

axillary emptying.

-Patients who agree to participate in the study.

Exclusion Criteria:

* Patients diagnosed with locally advanced breast cancer requiring extensive resection requiring reconstruction with extensive skin or myocutaneous flaps.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence of patients presenting seroma formation after mastectomy with or without axillary lymphadenectomy. | From enrollment to the end of treatment at 2 years
  -Number of patients presenting seroma after mastectomy with or without axillary lymphadenectomy in the case and control group.

SECONDARY OUTCOMES:
Time until the drain was removed after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  - Number of days until the drain is removed in the case and control group.
Amount of volume in the drains until it is removed after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  The number of millilitres in the drain until it is removed in the case and control group.
Time until seroma resolution after mastectomy with of without lymphadenectomy | From enrollment to the end of treatment at 2 years
  Number of days until resolution of the seroma in the case and control group.
Outpatient clinic visits after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  The number of outpatient clinic visits until the seroma is resolved in the case and control group.
Aspiration punctures after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  Number of aspiration punctures until the seroma is resolved in the case and control group.
Amount of punctures volume after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  The number of millilitres of all punctures performed until seroma resolution in the case and control group.
Emergency Department Visits after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  Number of visits to the emergency department due to seroma or drainage in the case and control group.
Types of complications after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  List of all the types of complications that occurred in the case and control group.
Incidence of complications after mastectomy with of without lymphadenectomy. | From enrollment to the end of treatment at 2 years
  Number of patients presenting each of the listed complications after surgery in the case and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egeli T, Sevinc AI, Bora S, Yakut MC, Cevizci T, Canda T, Sisman AR. Microporous polysaccharide hemospheres and seroma formation after mastectomy and axillary dissection in rats. Balkan Med J. 2012 Jun;29(2):179-83. doi: 10.5152/balkanmedj.2012.005. Epub 2012 Jun 1. PMID 25206991
- See also: Food and Drug Administration. Summary of safety and effectiveness — https://www.accessdata.fda.gov/cdrh_docs/pdf5/P050038b.pdf
- See also: BD. Arista™ AH Absorbable Hemostat — https://www.bd.com/en-us/products-and-solutions/products/product-families/arista-ah-absorbable-hemostat